CLINICAL TRIAL: NCT00584662
Title: Oxymetazoline Hydrochloride in Combination With Nasal Glucocorticosteroid for Perennial Allergic and Non-allergic Rhinitis in Subjects With Persistent Nasal Congestion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard Lockey, principal investigator, University of South Florida
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFRIN STUDY
Record Dates: First submitted 2007-12-21; First posted 2008-01-02 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2008-07

CONDITIONS: Chronic Rhinitis
Keywords: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Oxymetazoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Active Comparator): Oxymetazoline Hydrochloride
  Interventions: Drug: Oxymetazoline Hydrochloride

INTERVENTIONS:
Drug: Oxymetazoline Hydrochloride — Oxymetazoline Hydrochloride TWO SPRAYS BID
  Other Names: AFRIN

SUMMARY:
Nasal glucocorticosteroids (GCS) are considered first-line therapy for both allergic and non-allergic rhinitis.1-3 Nasal congestion can persist despite maximum treatment with intranasal GCS. No other drugs are superior to intranasal GCS in relieving nasal congestion. For example, antihistamines are not effective in relieving congestion.1 Oral decongestants are somewhat beneficial in relieving nasal congestion but can elevate blood pressure, cause restlessness, and cause urinary retention. Oxymetazoline, however, is a potent decongestant and the addition of it to a nasal GCS should add a considerable decongestant benefit. It may also be beneficial in patients with persistent nighttime congestion despite maximum dosages of nasal GCS.

Oxymetazoline is currently recommended for three days use because of the proposed risk of rhinitis medicamentosa,4 which is increased nasal congestion caused by prolonged use of nasal decongestant sprays.5-8 The term RM was coined early in the twentieth century after several case reports described patients developing rebound congestion after using first generation intranasal decongestants such as privine hydrochloride and ephedrine for prolonged periods6,7. The histopathology and mechanism of RM has been based on animal models which may not be pertinent to humans.9-13 Studies using oxymetazoline, a newer intranasal decongestant, in individuals without rhinitis have shown conflicting evidence for the development of RM.14-16 For example, normal individuals without rhinitis using oxymetazoline three times daily for four weeks did not develop RM.17 Also, it is unknown the frequency of administration and dosage of oxymetazoline it takes to induce RM or whether RM is just a return to a patient's baseline nasal congestion as present before beginning oxymetazoline. It is also unknown whether RM is more likely or only occurs with older vasoconstrictors such as privine hydrochloride and ephedrine rather than oxymetazoline.

Nasal GCS reduce the amount of rebound congestion in patients with perennial allergic rhinitis who have reportedly developed RM.18 Nasal GCS decrease nasal mucosa edema, recruitment of neutrophils and mononuclear cells, cytokine production, and late-phase nasal mediators.19-21 They may offer a protective benefit from the risk of developing RM. Oxymetazoline may also decrease inferior turbinate hypertrophy thereby permitting better adsorption of the nasal GCS.

Hypothesis

The addition of oxymetazoline to a nasal GCS for fourteen days will decrease the amount of congestion in subjects with allergic or non-allergic rhinitis with persistent congestion despite maximum recommended dosages of a nasal GCS. It is also hypothesized that nasal GCS protect against the development of RM secondary to oxymetazoline.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects 18 years of age and older
2. At least a one year history of perennial allergic or non-allergic rhinitis
3. Subjects receiving allergen immunotherapy must be on a stable maintenance regimen for at least 30 days before the first study visit and remain on this dosage during the study.
4. Subjects must be on the maximum doses of one of the following nasal GCS for at least one month: beclomethasone, flunisolide, fluticasone, mometasone, or triamcinolone.
5. Nasal Congestion Score of 2 or greater at screening visit (Day -7)
6. Average Nasal Congestion Score of 1.5 or greater at baseline visit (Day 1). Average Nasal Congestion Score is calculated from over the last three days prior to baseline and the morning of the baseline visit (i.e. total of seven scores)
7. Willingness to participate as indicated by signed informed consent

Exclusion Criteria:

1. Presence of hypersensitivity to oxymetazoline or mometasone
2. Women who are pregnant or lactating
3. Women of childbearing potential who are not abstinent or not practicing a medically acceptable form of contraception
4. Other nasal diseases likely to affect deposition of oxymetazoline such as sinusitis, nasal polyps, or nasal structural malformations
5. No respiratory tract infections in the last 14 days
6. Infections requiring antibiotics in the last 14 days
7. No oxymetazoline or other nasal sprays in the last 14 days
8. No cardiovascular disease, uncontrolled hypertension or hypertension requiring more than two drugs to achieve control, or arrythmias
9. Subjects can not be on beta or alpha blockers
10. No diabetes mellitus
11. No presence or history of ocular herpes simplex, cataracts, or glaucoma
12. Subjects who are currently alcohol or drug abusers
13. Inability to cooperate, comply with study procedures or communicate with the investigator as needed to successfully complete the study
14. No benign prostate hypertrophy
15. A history of psychosis
16. Patients with a planned hospitalization during the study
17. History of drug or alcohol abuse within the past five years
18. An infirmity, disability, or geographical location which seems likely to prevent regular attendance for patient visits
19. No use of the following medicines or therapies within the time period specified below prior to Day -7:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
to evaluate the effectiveness through symptom scores of the addition of oxymetazoline to nasal GCS in subjects with resistant congestion despite . | 9 WEEKS

SECONDARY OUTCOMES:
To evaluate the need for rescue medicine for persistent or worsening congestion.To evaluate evidence of rebound congestion in subjects treated with both nasal GCS and oxymetazoline.To evaluate improvement in the total nasal | 9 WEEKS

CONTACTS AND LOCATIONS:
Overall Officials: RICHARD F LOCKEY, MD, Principal Investigator — University of South Florida
Locations (1):
- USF, Tampa, Florida, United States